CLINICAL TRIAL: NCT01889654
Title: Analysis of Frequency and Phenotype of Anti-nucleosome B Lymphocyte in Systemic Lupus
Brief Title: Anti-nucleosome B Lymphocytes in Lupus
Status: Terminated | Type: Observational
Why Stopped: recrutment difficulty
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5543
Record Dates: First submitted 2013-06-25; First posted 2013-06-28 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-01

CONDITIONS: Systemic Lupus Erythematosus With or Without Clinical Activity
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (2):
- patient
  Interventions: Other: Venous blood sampling
- healthy volunteers
  Interventions: Other: Venous blood sampling

INTERVENTIONS:
Other: Venous blood sampling

SUMMARY:
Lupus disease is characterized by the production of pathogenic autoantibodies, which participate in end-organ damages. The phenotype of B cells producing the pathogenic autoantibodies in lupus patients is today unknown. Antinucleosome antibodies are characteristic of lupus disease.This project proposes to detect antinucleosome B cells in lupus patients and to analyse their phenotype and their frequency.

ELIGIBILITY:
Inclusion criteria for SLE patients:

SLE patient : diagnostic based on ACR criteria

* SLE patient producing seric anti-nucleosome antibodies (ELISA)
* SLEDAI-2K activity score : inferior to 5 for quiescent patients, superior to 8 since at least 2 months for active patients

Exclusion criteria for SLE patients:

-- Other autoimmune diseases than SLE- Induced lupus

* Treatment with corticosteroids >10mg/d (prednisone) for quiescent patients
* Treatment with corticosteroids >20mg/d (prednisone) for active patients
* Oral immunosuppressive treatment during the last 6 months (methotrexate, azathioprine, ciclosporine, mycophénolate mofétil) for all patients, treatment during the last year with cyclophosphamide or monoclonal antibodies (rituximab, belimumab) for pour quiescent patients
* Disease which can modify B and T lymphocyte functions: primary immune deficiencies, evolutive infections, chronic viral infection (VIH in particular), chemotherapy or neoplasm antecedent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: lupus patient and healthy volunteers
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
all cause mortality | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, Bas Rhin, France